CLINICAL TRIAL: NCT00181636
Title: Galantamine-CR and Cognitive Dysfunction in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003P-000030/24
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Galantamine-CR

SUMMARY:
The purpose of the study is to determine whether the investigational drug galantamine-CR (Reminyl- Controlled Release capsule) is useful in improving problems with memory in bipolar patients with stable mood. This study is being done because a large proportion of patients with bipolar disorder experience significant memory problems, even when their mood is stable, after adequate treatment. These memory problems have been associated with poor daily social functioning. Studying galantamine-CR in this population may provide a new clinical way to combat memory problems in stable patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnostic criteria for bipolar disorder
* men or women aged 18-65
* a baseline Hamilton-D17 score of < 10 at screen visit
* a baseline YMRS score of < 10 at screen visit
* no acute episodes of depression or mania for the previous 12 weeks.
* written informed consent

Exclusion Criteria:

* Subjects with current suicidal ideation
* Pregnant women or women of childbearing potential
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease; History of seizure disorder, brain injury, any history of known neurological disease (multiple sclerosis, degenerative disease such as ALS, Parkinson disease and any movement disorders, etc)
* History or current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, major depressive disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 12 months
* History of multiple adverse drug reactions
* Patients with mood congruent or mood incongruent psychotic features Subjects who are active smokers or who stopped smoking less than 3 months prior to enrollment; Clinical or laboratory evidence of hypothyroidism
* Patients who have had an episode of acute depression or mania during the 12 weeks prior to enrollment
* Patients who have had electroconvulsive therapy (ECT) within the 6 months preceding enrollment
* Patients with physical contraindications to magnetic resonance spectroscopy (ferrous surgical clips, cardiac pacemakers, ferrous prosthesis)
* Patients taking any of the following medications: other cholinesterase inhibitors, succinylcholine, neuromuscular blocking agents, cholinergic agonists (e.g., bethanechol), cimetidine, ketoconazole, erythromycin, fluoxetine, paroxetine, and fluvoxamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
neurocognitive testing at last study visit (18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Dan V Iosifescu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Bipolar Clinic and Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Iosifescu DV, Moore CM, Deckersbach T, Tilley CA, Ostacher MJ, Sachs GS, Nierenberg AA. Galantamine-ER for cognitive dysfunction in bipolar disorder and correlation with hippocampal neuronal viability: a proof-of-concept study. CNS Neurosci Ther. 2009 Winter;15(4):309-19. doi: 10.1111/j.1755-5949.2009.00090.x. PMID 19889129